CLINICAL TRIAL: NCT05498168
Title: Computational Prediction and Experimental Validation of Esophageal Cancer Associated Neoantigens
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 61/GCN-HDDD
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Cancer; Neoantigen
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: ratio of predicted neoantigens — 10 ml of whole blood is collected from each patient prior surgery Fresh tumor tissue samples (~ 1cm3 ) are collected during surgery

SUMMARY:
This study is to develop computational pipelines and experimental validation assays for improving the identification of neoantigens from patients with esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the common malignant tumor with poor survival. The long-term surival rate of patients with advanced EC stages has not been improved with multidisciplinary treatments including surgery and chemotherapy and radiation. Recently, immunotherapy approaches using checkpoint inhibitors (CPI), cancer vaccine, and adoptive T cell therapy have improved survival outcomes of EC patients. The clinical outcomes are associated with expression levels as well as the immunogenicity of neoantigens which arise from soma mutations. Therefore, the identification of immunogenic neoantigens is essential for achieving effective therapies. Recent data published by the Tumor Neoantigen Selection Alliance (TESLA) show that the majority (98%) of predicted neoantigens are lack of immunogenicity and ineffective in activating antitumor immune responses. In our study, we aim to develop a pipeline with both computational prediction tools and experimental validation assays to enhance the accuracy of neoantigen identification.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged 18 years and older
2. Diagnosed with advanced esophageal cancer
3. Treatment-Naive
4. Not known for other concomitant cancers
5. Provide written informed consent

Exclusion Criteria:

1. Insufficient tumor tissues (less than 1 cm3 )
2. Unable to sign informed consent
3. Underwent treatment

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who were diagnosed with adavanced esophageal cancer and underwent surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The neoantigen landscape of patients with esophageal cancer | 3 months from the begining of study
  The analysis of tumor DNA and RNA sequencing data will provide the mutational distribution of patients with esophageal cancer, which could give rise to neoantigens. Of those, neoantigens derived from hotspot mutations in Vietnamese esophageal cancer patients will be identified.
The ratio of predicted neoantigens being presented by HLA-I | 6 months from the begining of study
  Computational pipelines will be employed to predict the pairing of neoantigens and HLA molecules. Subsequently, the ratio of those predicted neoantigens will be validated by co-immunoprecipitation with anti-HLA antibodies and mass spectrometry analysis for their binding to corresponding HLA molecules.
The ratio of predicted neoantigens being immunogenic | 12 months from the begining of study
  Immunoassays will be employed to identify neoantigens that could activate CD4 and CD8 T cells to kill tumor cells and serve as putative candidates for immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No